CLINICAL TRIAL: NCT04875598
Title: COMPARISON OF LAPAROSCOPY AND ULTRASOUND ASSISTED TRANSVERSUS ABDOMINIS PLANE BLOCK METHODS IN LAPAROSCOPIC TOTAL EXTRAPERITONEAL HERNIA REPAIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, MD. Anil Ergin, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: drANILERGIN
Record Dates: First submitted 2021-05-01; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain; Inguinal Hernia; Transversus Abdominis Plane Block
Keywords: inguinal hernia; Transversus abdominis plane block; postoperative pain; Total extraperitoneal hernia repair
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: A total of 60 patients will be included in the study; Group 1: 30 patients will be injected with local anesthetic into the fascia between the transversus abdominis and internal oblique muscles with the help of ultrasound from the designated area (Before the operation starts, TAPBwith 20 ml 0.25 % bupivacaine will be applied to the surgical side under ultrasonography)
  Group 2: 30 patients, local anesthetic injection will be made to the same area under laparoscopic direct vision. 50 mg Bupivacaine (0.25 % 20 ml bupivacaine solution) has been determined as the application dose and this amount will be applied in both groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): 30 patients will be injected with local anesthetic into the fascia between the transversus abdominis and internal oblique muscles with the help of ultrasound from the designated area (Before the operation starts, TAPBwith 20 ml 0.25 % bupivacaine will be applied to the surgical side under ultrasonography)
  Interventions: Procedure: Ultrasound assisted - Laparoscopy assisted Transversus Abdominis Plane Block
- Group 2 (Active Comparator): 30 patients, local anesthetic injection will be made to the same area under laparoscopic direct vision. 50 mg Bupivacaine (0.25 % 20 ml bupivacaine solution) has been determined as the application dose and this amount will be applied in both groups.
  Interventions: Procedure: Ultrasound assisted - Laparoscopy assisted Transversus Abdominis Plane Block

INTERVENTIONS:
Procedure: Ultrasound assisted - Laparoscopy assisted Transversus Abdominis Plane Block — Ultrasound assisted TAPB application will be applied by an anesthesiology and reanimation specialist and Laparoscopy assisted TAPB application will be applied by the surgeon performing the operation.

SUMMARY:
While the rate of inguinal hernia repair operations in England is 10 per 100,000 people. The rate in the United States is found to be 28 per 100,000 people. Today, the effectiveness between open repair and laparoscopic repair in inguinal hernia repair is still debated. Laparoscopic approach offers many advantages over open repair. Regional blocks have an important place in the multi-modal anesthesia approach applied to reduce postoperative pain. In this sense, the Transversus Abdominis Plane Block (TAPB) emerges as an effective regional anesthesia method that reduces postoperative pain. This method can be applied with the help of ultrasound or laparoscopy. The aim of this study is to compare the ultrasound-assisted TAPB application and Laparoscopy-assisted TAPB application in Total Extraperitoneal hernia repair (TEP) to reveal the effects of postoperative pain.

A total of 60 patients will be included in the study; 30 of these patients will be injected with local anesthetic into the fascia between the transversus abdominis and internal oblique muscles with the help of ultrasound from the designated area (Before the operation starts, TAPB with 20 ml 0.25 % bupivacaine will be applied to the surgical side under ultrasonography); In the other 30 patients, local anesthetic injection will be made to the same area under laparoscopic direct vision. 50 mg Bupivacaine (0.25 % 20 ml bupivacaine solution) has been determined as the application dose and this amount will be applied in both groups.

10 cm visual analog scale (VAS) will be used in postoperative pain follow-up. 50 mg intravenous tramadol will be administered to patients with VAS > 4 and tramadol will be supplemented to 100 mg in patients with high pain levels after 30 minutes. Oral non-steroidal anti-inflammatory will be given at the postoperative 8th hour. Patients whose pain persists despite current therapy will be given 25 mg of meperidine intravenously as a rescue analgesic. The doses of analgesic administered in the postoperative period and the hours of administration will be recorded

DETAILED DESCRIPTION:
While the rate of inguinal hernia repair operations in England is 10 per 100,000 people. The rate in the United States is found to be 28 per 100,000 people. Today, the effectiveness between open repair and laparoscopic repair in inguinal hernia repair is still debated. Laparoscopic approach offers many advantages over open repair. These are topics such as postoperative pain, quick recovery, and shortening of returning to work. Postoperative pain is the most important determinant of recovery after abdominal surgeries. Postoperative pain can be explained by two pathways connected to the peritoneum; The first is the parietal peritoneum, which has a very rich innervation, and the other is the visceral peritoneum stimulated by the vagus. In order to eliminate these peritoneal pains, surgeons have been injecting local anesthetic into various areas on the anterior abdominal wall and intraperitoneal space since 1950. Regional blocks have an important place in the multi-modal anesthesia approach applied to reduce postoperative pain. In this sense, the Transversus Abdominis Plane Block (TAPB) emerges as an effective regional anesthesia method that reduces postoperative pain. TAPB; It is a type of regional anesthesia applied to the facial plane between the internal oblique muscle and the transversus abdominis muscles, targeting the somatic nerves (T6 - L1). This method can be applied with the help of ultrasound or laparoscopy. The aim of this study is to compare the ultrasound-assisted TAPB application and Laparoscopy-assisted TAPB application in Total Extraperitoneal hernia repair (TEP) to reveal the effects of postoperative pain.

TEP will be performed with 2-3 mg / kg propofol, 2 mcg / kg fentanyl and 0.6 mg / kg rocuronium in patients who will undergo anesthesia induction with BIS < 60, after intubation, 40 % oxygen / 1.5 - 2 % sevoflurane inhalation will be applied to keep the BIS value between 40 - 60 in 60 % air. Before the operation starts, TAPB will be made with 20 ml 0.25 % bupivacaine in the direction of ultrasonography on the side to be operated. During the operation, if there is a 20 % increase in blood pressure and heart rate from baseline, 0.5 mcg / kg intravenous fentanyl will be administered and the administered fentanyl dose will be recorded. 1gr paracetamol 30 minutes before the end of the operation and 4 mg ondansetron 15 minutes before the end of the operation will be administered intravenously. With the help of a 22 G injector, local anesthetic injection will be made from the anterior to the area where the midaxillary line intersects the Bogros area. Digital examination will be performed to define the injection site and the injection area will be determined.

A total of 60 patients will be included in the study; 30 of these patients will be injected with local anesthetic into the fascia between the transversus abdominis and internal oblique muscles with the help of ultrasound from the designated area (Before the operation starts, TAPB with 20 ml 0.25 % bupivacaine will be applied to the surgical side under ultrasonography); In the other 30 patients, local anesthetic injection will be made to the same area under laparoscopic direct vision. 50 mg Bupivacaine (0.25 % 20 ml bupivacaine solution) has been determined as the application dose and this amount will be applied in both groups. Bart 3D anatomical polypropylene patch will be used in both groups and the patch will be attached with the help of 1 absorbable tacker. Carbon dioxide gas will be given to the preperitoneal area at a rate of 4 - 6 L / min and at a pressure of 15 mm Hg. 3 trocars will be used; One 10 mm camera trocar and two 5 mm working trocars will be entered through the midline below the navel. At the end of the operation, the patients will be extubated by antagonizing the muscle relaxant effect with 0.02 mg / kg atropine and 0.05 mg / kg neostigmine. 10 cm visual analog scale (VAS) will be used in postoperative pain follow-up. 50 mg intravenous tramadol will be administered to patients with VAS > 4 and tramadol will be supplemented to 100 mg in patients with high pain levels after 30 minutes. Oral non-steroidal anti-inflammatory will be given at the postoperative 8th hour. Patients whose pain persists despite current therapy will be given 25 mg of meperidine intravenously as a rescue analgesic. The doses of analgesic administered in the postoperative period and the hours of administration will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Patients who underwent total extraperitoneal hernia repair
* Patients without any postoperative complications
* Patients who cannot be drained for any reason

Exclusion Criteria:

* Patients who underwent another hernia repair technique during surgery for any reason.
* Patients who do not want to participate in the study
* Patients with any complications after surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours
  10 cm visual analog scale (VAS) will be used in postoperative pain follow-up. 10: too much pain , 1: no pain

SECONDARY OUTCOMES:
patient satisfaction | 24 hours
  Patients will be evaluated with a patient satisfaction questionnaire after surgery. 5: Very satisfied , 1:Not satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih sultan mehmet training and research hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided